CLINICAL TRIAL: NCT05600127
Title: Chemotherapy and Sequential Immunotherapy for Locally Advanced Urothelial Cancer: the CHASIT Study
Brief Title: Chemotherapy and Sequential Immunotherapy for Locally Advanced Urothelial Cancer
Acronym: CHASIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, J.L. Boormans, MD PhD, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL80678.078.22
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Urothelial Carcinoma
Keywords: Chemotherapy; Immunotherapy; Safety; Pathological response
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Masking Description: single arm study, therefore no masking possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab (Experimental): 3 cycles of avelumab (Bavencio), 800mg intravenous instillation in 60 min, every 2 weeks.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — 3 cycles of avelumab (800mg, every 2 weeks)
  Other Names: Bavencio

SUMMARY:
Patients with locally advanced or clinically node positive urothelial carcinoma treated with chemotherapy, will receive 3 cycles of avelumab, followed by radical surgery.

DETAILED DESCRIPTION:
Patients with locally advanced or clinically node positive urothelial carcinoma of the bladder, ureter or urethra (cT4NxM0 or cTxN1-N3M0) with at least stable disease after treatment with 3-4 cycles of platinum-based chemotherapy, will be treated with 3 cycles of avelumab (anti-PD-L1). If there are no signs of disease progression after avelumab treatment, radical surgery of the primary tumor and a pelvic lymph node dissection will follow.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Have histologically confirmed urothelial carcinoma of the bladder, upper urinary tract or urethra; a maximum of 50% of aberrant histology is allowed.
3. Have clinical stage cT4NxM0 or cTxN1-N3M0 as assessed by bimanual examination under anaesthesia, CT scan, MRI scan or PET-CT scan.
4. Have at least stable disease after a minimum of 3 or a maximum of 4 cycles of induction chemotherapy with cisplatin / carboplatin + gemcitabine according to RECIST v1.1.
5. Are fit and willing to undergo radical surgery with removal of lymph node template including all affected lymph nodes and the primary tumor.
6. World Health Organisation performance status of 0-2.
7. Provide written informed consent.
8. Negative pregnancy test in women with childbearing potential.
9. Adequate bone marrow function, including:

   1. Absolute neutrophil count (ANC) ≥1,500/mm3 or 1.5 x 109/L;
   2. Platelets ≥100 x 109/L;
   3. Hemoglobin ≥5.6 mmol/L (may have been transfused).
10. Adequate renal function, defined as estimated creatinine clearance ≥30 mL/min as calculated by the CKD-EPI eGFR.
11. Adequate liver function, including:

    1. Total serum bilirubin <1.5 x upper limit of normal (ULN);
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x ULN.

Exclusion Criteria:

1. Predominant (>50%) non-urothelial carcinoma histology in the diagnostic endoresection specimen of the bladder, urethra or upper urinary tract.
2. Any test for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection.
3. Have an estimated creatinin clearance as assessed by the CKD-EPI eGFR of <30 ml/min.
4. Prior exposure to immune-mediated therapy with exclusion of Bacillus-Calmette Guérin intravesical instillations, including but not limited to other anti-CTLA-4, anti PD-1, anti PD-L1, or anti-PD-L2 antibodies.
5. Persisting toxicity related to prior chemotherapy (Grade >2 NCI CTCAE v5.0).
6. A diagnosis of any other malignancy within 2 years prior to inclusion, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the breast or of the cervix, low grade prostate cancer on surveillance without any plans for treatment intervention, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease.
7. ≤2 cycles of induction platinum-based chemotherapy received.
8. Progression of disease during or following induction platinum-based chemotherapy, as assessed by RECIST v1.1.
9. Distant metastatic disease.
10. Previous pelvic radiation therapy.
11. Breastfeeding women.
12. Bilateral upper urinary tract urothelial carcinoma.
13. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
14. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
15. Active infection requiring systemic therapy.
16. Known severe hypersensitivity reactions to monoclonal antibodies (Grade 3), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of asthma symptom control per the Global Initiative for Asthma 2015).
17. Known prior or suspected hypersensitivity to avelumab.
18. Current use of immunosuppressive medication, EXCEPT the following:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
    2. Systemic corticosteroids at (equivalent) doses of maximum 10 mg prednisone;
    3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
19. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy, or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
20. Vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivate vaccines (for example, inactivated influenza vaccines) or mRNA vaccines (for example, COVID-19 vaccines).
21. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, and pneumonitis; psychiatric condition including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | About 1 month after radical surgery
  the proportion of patients without residual UC in the surgical resection specimen, ypT0N0 (carcinoma situ is allowed), in the intention-to-treat analysis.

SECONDARY OUTCOMES:
Survival | 24 months after radical surgery
  Progression-free, cancer-specific and overall survival at 24 months, calculated from the time of 1st administration of avelumab
Adverse events | 90 days after administration of the last cycle of avelumab
  Adverse events of assessed by the CTCAE v5.0
Surgical complications | 90 days after radical surgery
  Assesed by Clavien-Dindo classification within 30 and 90 days from date of surgery
Non-invasive urothelial cancer | About 1 month after radical surgery
  The rate of non-invasive urothelial cancer in the surgical resection specimen, stage ypT0N0/ypTisN0/ypTaN0/ypT1N0
Delay in surgery | About 1 month after radical surgery
  The proportion of patients in whom radical surgery is delayed >8 weeks after last administration of avelumab due to toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: J L Boormans, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - Radboud UMC, Nijmegen, Gelderland
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Amphia ziekenhuis, Breda, North Brabant
  - Erasmus MC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutten VC, Salhi Y, Robbrecht GJ, de Wit R, van Leenders GJLH, Zuiverloon TCM, Boormans JL. The CHASIT study: sequential chemo-immunotherapy in patients with locally advanced urothelial cancer - a non-randomized phase II clinical trial. BMC Cancer. 2023 Jun 13;23(1):539. doi: 10.1186/s12885-023-10963-7. PMID 37312054